CLINICAL TRIAL: NCT04154982
Title: Cardiac Arrhythmia Catheter Ablation Procedures Guided by x-Ray Imaging: N-Acetylcysteine Protection Against Radiation Induced Cellular damagE (CARAPACE Study)
Brief Title: N-Acetylcysteine Protection Against Radiation Induced Cellular Damage
Acronym: CARAPACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Principal Investigator, Claudio Tondo, Deputy of Heart Rhythm Center, Centro Cardiologico Monzino
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCM1006
Record Dates: First submitted 2019-10-17; First posted 2019-11-07 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cardiac Arrhythmia
Keywords: Electrophysiology; Arrhythmias; Arrhythmia ablation; Ionizing radiation risk; Oxidative stress; DNA damage biomarkers
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Researchers, involved in the assessment of NAC efficacy, are blinded to randomization process; thus, they do not know whether the patients are in the NAC or in the control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmacological treatment (Experimental): Patients are treated with NAC prior to carrying out CAP.
  Interventions: Drug: Acetyl cysteine
- Standard procedure (No Intervention): Patients are not treated with NAC. No placebo treatment is performed.

INTERVENTIONS:
Drug: Acetyl cysteine — 1200 mg of NAC are intravenously administrated 1 hour prior to carrying out CAP.
  Arms: Pharmacological treatment

SUMMARY:
Catheter ablation procedures (CAPs) are first line treatment for a great variety of cardiac arrhythmias. CAPs require X-Ray imaging; consequently, CAPs cause ionizing radiation (IR) exposure for patients. Exposure to IR, even at low-doses, increases individual risk of developing cancer. IR cause DNA damage directly and, mostly, indirectly by formation of cellular free radicals. Furthermore different response to IR results from inherited variants in genes involved in DNA damage repair. N-acetylcysteine (NAC) is an aminoacid that can directly neutralize free radicals and increase antioxidant systems. Our preliminary data suggest that IR exposure in patients undergoing CAP deranges the oxidative stress status and the pre-procedure intravenous administration of NAC could decrease such abnormality.

DETAILED DESCRIPTION:
CARAPACE is a prospective, randomized, single-blinded, parallel-arm monocenter study. Eligible patients undergoing CAP at the Arrhythmology Unit of Centro Cardiologico Monzino will be enrolled.

The hypothesis driving our study, based on published literature and our preliminary data, is that administration of antioxidant agents, before cardiac procedures involving IR exposure, might prevent IR harmful effects on human tissues in terms of reduction of systemic oxidative stress status and, in parallel, of oxidative DNA damage.

The antioxidant agent tested in our study is NAC. NAC is a well-tolerated and safe medication and it has antioxidant properties is based on three main mechanisms: 1) direct antioxidant effect, 2) glutathione (GSH) precursor action, and 3) its activity in breaking thiolated proteins.

Another hypothesis to be tested is whether genes involved in DNA damage repair could explain the great variability in patient radiosensitivity to IR exposure and whether these genes could affect NAC protective/healing effects.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age >18 years.
* Negative hCG pregnancy test (if appropriate).
* Indication to perform CAP guided by fluoroscopy (IR imaging).
* Ability and willingness to give informed consent and to comply with protocol.

Exclusion Criteria:

* Any contraindication to CAP (such as, pregnancy and breastfeeding).
* Hypersensitivity to the active substance or to any of the excipients.
* Enrollment in another study that may interfere with CARAPACE study.
* Administration of an experimental drug within 30 days or 5 half-lives of the investigational drug.
* Chronic kidney disease (serum creatinine >1.5 mg/dl).
* Acute/Chronic inflammatory disease.
* Antioxidant drugs intake over the previous 2 weeks.
* History of radiotherapy or chemotherapy in the last year.
* Any documented condition that, in PI's motivated judgement, makes the patient a poor candidate for the study.
* Computed tomography and/or coronary angiography within 5 days prior to baseline analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Measurement of change in systemic oxidative stress (ratio between GSH oxidized form (GSSG) and GSH, 8-iso-prostaglandinF2α (8-iso-PGF2α) and 8-hydroxy-2-deoxyguanosine (8-OHdG)) and genomic DNA oxidative damage (percentage of DNA present in the tails). | 48 hours
  Measurement of change in systemic oxidative stress (GSSG/GSH, 8-iso-PGF2α and 8-OHdG) and genomic DNA oxidative damage (% DNA present in the tails of the comet assay) between the two groups (NAC versus no NAC) at the different time-points (T0 = before CAP, T1 = 3h after CAP, T2 = 24h after CAP, T3 = 48h after CAP).

SECONDARY OUTCOMES:
Measurement of change in systemic oxidative stress (GSSG/GSH, 8-iso-PGF2α and 8-OHdG) and genomic DNA oxidative damage (% DNA present in the tails) related to IR dose (fluoroscopy time (FT), Dose Area Product (DAP) and effective dose (ED)). | 48 hours
  Measurement of change in systemic oxidative stress (GSSG/GSH, 8-iso-PGF2α and 8-OHdG) and genomic DNA oxidative damage (% DNA present in the tails) related to IR dose (FT, DAP and ED) between the two groups (NAC versus no NAC).
Measurement of change in genomic DNA oxidative damage (% DNA present in the tails) related to IR dose (FT, DAP and ED) and inherited variants in genes involved in DNA damage repair. | 48 hours
  Measurement of change in genomic DNA oxidative damage (% DNA present in the tails) related to IR dose (FT, DAP and ED) and inherited variants in genes involved in DNA damage repair between the two groups (NAC versus no NAC).
Measurement of change in the response to NAC administration related to inherited variants in genes involved in DNA damage repair. | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Cardiologico Monzino, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turnu L, Porro B, Alfieri V, Di Minno A, Russo E, Barbieri S, Bonomi A, Dello Russo A, Tondo C, D'Alessandra Y, Cavalca V, Tremoli E, Colombo GI, Casella M. Does Fluoroscopy Induce DNA Oxidative Damage in Patients Undergoing Catheter Ablation? Antioxid Redox Signal. 2018 Apr 20;28(12):1137-1143. doi: 10.1089/ars.2017.7334. Epub 2017 Nov 27. PMID 28938845
- [Background] Heidbuchel H, Wittkampf FH, Vano E, Ernst S, Schilling R, Picano E, Mont L, Jais P, de Bono J, Piorkowski C, Saad E, Femenia F. Practical ways to reduce radiation dose for patients and staff during device implantations and electrophysiological procedures. Europace. 2014 Jul;16(7):946-64. doi: 10.1093/europace/eut409. Epub 2014 May 2. PMID 24792380
- [Background] Evans MD, Dizdaroglu M, Cooke MS. Oxidative DNA damage and disease: induction, repair and significance. Mutat Res. 2004 Sep;567(1):1-61. doi: 10.1016/j.mrrev.2003.11.001. PMID 15341901
- [Background] Andreassi MG, Foffa I, Manfredi S, Botto N, Cioppa A, Picano E. Genetic polymorphisms in XRCC1, OGG1, APE1 and XRCC3 DNA repair genes, ionizing radiation exposure and chromosomal DNA damage in interventional cardiologists. Mutat Res. 2009 Jun 18;666(1-2):57-63. doi: 10.1016/j.mrfmmm.2009.04.003. Epub 2009 Apr 22. PMID 19393248
- [Background] Huang A, Glick SA. Genetic susceptibility to cutaneous radiation injury. Arch Dermatol Res. 2017 Jan;309(1):1-10. doi: 10.1007/s00403-016-1702-3. Epub 2016 Nov 22. PMID 27878387
- [Background] Cervelli T, Panetta D, Navarra T, Gadhiri S, Salvadori P, Galli A, Caramella D, Basta G, Picano E, Del Turco S. A New Natural Antioxidant Mixture Protects against Oxidative and DNA Damage in Endothelial Cell Exposed to Low-Dose Irradiation. Oxid Med Cell Longev. 2017;2017:9085947. doi: 10.1155/2017/9085947. Epub 2017 Aug 9. PMID 28852434
- [Background] Aldini G, Altomare A, Baron G, Vistoli G, Carini M, Borsani L, Sergio F. N-Acetylcysteine as an antioxidant and disulphide breaking agent: the reasons why. Free Radic Res. 2018 Jul;52(7):751-762. doi: 10.1080/10715762.2018.1468564. Epub 2018 May 9. PMID 29742938
- [Background] Mu H, Sun J, Li L, Yin J, Hu N, Zhao W, Ding D, Yi L. Ionizing radiation exposure: hazards, prevention, and biomarker screening. Environ Sci Pollut Res Int. 2018 Jun;25(16):15294-15306. doi: 10.1007/s11356-018-2097-9. Epub 2018 Apr 29. PMID 29705904
- [Background] Squellerio I, Caruso D, Porro B, Veglia F, Tremoli E, Cavalca V. Direct glutathione quantification in human blood by LC-MS/MS: comparison with HPLC with electrochemical detection. J Pharm Biomed Anal. 2012 Dec;71:111-8. doi: 10.1016/j.jpba.2012.08.013. Epub 2012 Aug 23. PMID 22947504
- [Background] Turnu L, Di Minno A, Porro B, Squellerio I, Bonomi A, Manega CM, Werba JP, Parolari A, Tremoli E, Cavalca V. Assessing Free-Radical-Mediated DNA Damage during Cardiac Surgery: 8-Oxo-7,8-dihydro-2'-deoxyguanosine as a Putative Biomarker. Oxid Med Cell Longev. 2017;2017:9715898. doi: 10.1155/2017/9715898. Epub 2017 Jun 4. PMID 28660009
- [Background] Cavalca V, Minardi F, Scurati S, Guidugli F, Squellerio I, Veglia F, Dainese L, Guarino A, Tremoli E, Caruso D. Simultaneous quantification of 8-iso-prostaglandin-F(2alpha) and 11-dehydro thromboxane B(2) in human urine by liquid chromatography-tandem mass spectrometry. Anal Biochem. 2010 Feb 15;397(2):168-74. doi: 10.1016/j.ab.2009.10.014. Epub 2009 Oct 13. PMID 19825360
- [Background] Purcell S, Neale B, Todd-Brown K, Thomas L, Ferreira MA, Bender D, Maller J, Sklar P, de Bakker PI, Daly MJ, Sham PC. PLINK: a tool set for whole-genome association and population-based linkage analyses. Am J Hum Genet. 2007 Sep;81(3):559-75. doi: 10.1086/519795. Epub 2007 Jul 25. PMID 17701901
- [Background] Amadio P, Colombo GI, Tarantino E, Gianellini S, Ieraci A, Brioschi M, Banfi C, Werba JP, Parolari A, Lee FS, Tremoli E, Barbieri SS. BDNFVal66met polymorphism: a potential bridge between depression and thrombosis. Eur Heart J. 2017 May 7;38(18):1426-1435. doi: 10.1093/eurheartj/ehv655. PMID 26705390
- [Background] Casella M, Dello Russo A, Russo E, Catto V, Pizzamiglio F, Zucchetti M, Majocchi B, Riva S, Vettor G, Dessanai MA, Fassini G, Moltrasio M, Tundo F, Vignati C, Conti S, Bonomi A, Carbucicchio C, Di Biase L, Natale A, Tondo C. X-Ray Exposure in Cardiac Electrophysiology: A Retrospective Analysis in 8150 Patients Over 7 Years of Activity in a Modern, Large-Volume Laboratory. J Am Heart Assoc. 2018 May 22;7(11):e008233. doi: 10.1161/JAHA.117.008233. PMID 29789334
- [Background] Catto V, Stronati G, Porro B, Fiorelli S, Ricci V, Vavassori C, Russo E, Guerra F, Gasperetti A, Ribatti V, Sicuso R, Dello Russo A, Veglia F, Tondo C, Cavalca V, Colombo GI, Tremoli E, Casella M. Cardiac arrhythmia catheter ablation procedures guided by x-ray imaging: N-acetylcysteine protection against radiation-induced cellular damage (CARAPACE study): study design. J Interv Card Electrophysiol. 2021 Sep;61(3):577-582. doi: 10.1007/s10840-020-00853-4. Epub 2020 Aug 24. PMID 32833109
- See also: Expert Consensus Document on Optimal Use of Ionizing Radiation in Cardiovascular Imaging — http://doi.org/10.1016/j.jacc.2018.02.017
- See also: National Research Council. 2006. Health Risks from Exposure to Low Levels of Ionizing Radiation: BEIR VII Phase 2. Washington, DC: The National Academies Press. — http://doi.org/10.17226/11340